## **GEINO-13**

Phase II pilot, open, multicenter and prospective clinical trial to evaluate the safety and efficacy of Palbociclib (PD0332991), an inhibitor of cyclin-dependent kinases 4 and 6 (CDK4 and CDK6), in patients with recurrent Oligodendroglioma with preservation of the activity of the RB protein

# FINAL STATISTICAL REPORT TABLES, LISTS AND FIGURES



xxth of xxxxxxx de xxxx (version xx)

### SPONSOR

### STUDY CHIEF INVESTIGATOR

### MONITORING ORGANISATION (CRO)

DATE: 29/11/2022 (version 1.3)

### **INDEX**

| ••• | | =7: | |
|---|---|---|---|
| <u>1.</u> | RI | ESULTS (TABLES, LISTS AND FIGURES) | 6 |
| | <u>1.1.</u> | STUDY POPULATION | 6 |
| | | 1.1.1. SCREENED PATIENTS | 6 |
| | <u>1.2.</u> | DEMOGRAPHIC AND CLINICAL BASELINE CHARACTERISTICS | 8 |
| | | 1.2.1. CLINICAL BASELINE CHARACTERISTICS | 8 |
| | | 1.2.2. CLINICAL TUMOUR CHARACTERISTICS | 9 |
| | | 1.2.3. PREVIOUS PATHOLOGIES | 13 |
| | <u>1.3.</u> | EFFICACY ANALYSES | 17 |
| | | 1.3.1. PRIMARY EFFICACY ANALYSES: PFS | 17 |
| | | 1.3.2. SECONDARY EFFICACY ANALYSES | 19 |
| | <u>1.4.</u> | SAFETY ANALYSES | 32 |
| | | 1.4.1. ADEVERSE EVENTS | 32 |
| | | 1.4.2. TOXICITIES | 35 |
| | | 1.4.3. SERIOUS ADVERSE EVENTS | 37 |
| | <u>1.5.</u> | ANNEX I: LIST OF ALL TOXICITIES | 38 |
| | <u>1.6.</u> | ANNEX II: ADDITIONAL RESULTS | 41 |
| | | 1.6.1. LONG SURVIVORS | 41 |
| | | $\underline{\textbf{1.6.2.}} \ \underline{\textbf{BASELINE}} \ \underline{\textbf{AND}} \ \underline{\textbf{TUMOUR}} \ \underline{\textbf{CHARACTERISTICS}} \ \underline{\textbf{VS}} \ \underline{\textbf{LONG}} \ \underline{\textbf{SURVIVORS}}$ | 42 |
| | | 1.6.3 ADDITIONAL FIGURES | 43 |

DATE: 29/11/2022 (version 1.3)


### **Tables:**

| <u>Table 1. Screened patients</u> | 6 |
|---|---|
| Table 2. Evaluable patients | 6 |
| Table 3. Patients included and excluded from each hospital | 6 |
| Table 4. List of patients excluded from the analysis | 7 |
| Table 5. Age | 8 |
| Table 6. Gender and race | 8 |
| Table 7. Clinical data | 8 |
| Table 8. Analytical data | 8 |
| Table 9. Biochemistry data | 8 |
| Table 10. Coagulation data | 9 |
| Table 11. Thyroid function | 9 |
| Table 12. ECG | 9 |
| Table 13. First surgery characteristics | 9 |
| Table 14. List of patients with diagnosisin first surgery | 10 |
| Table 15. Last surgery characteristics | 11 |
| Table 16. Deletion | 11 |
| Table 17. Surgery compliance | 12 |
| Table 18. Baseline Barthel Index and Minimental test | 12 |
| Table 19. Previous pathologies | 13 |
| Table 20. List of previous pathologies | 15 |
| Table 21. Time since diagnosis | 16 |
| Table 22. Progression Free Survival | 17 |
| Table 23. Time until PD/exitus (only pts with event) | 18 |
| Table 24. Overall Survival | 19 |
| Table 25. Time until exitus (only deaths) | 20 |
| Table 26. Time of follow-up (all patients) | 20 |
| Table 27. Best response and Clinical benefit rate | 21 |
| Table 28. Status at end of study | 21 |
| Table 29. RANO Evaluation (I) | 22 |
| Table 30. RANO Evaluation (II) | 23 |
| Table 31. List of patients with RANO progressions with deatils | 24 |
| Table 32. Use of Corticoids | 25 |
| Table 33. List of patients receiving corticoids and Follow-up of dosage | 25 |
| Table 34. Minimental Test: Results for each patient | 26 |
| Table 35. Minimental Test: Summary in each visit | 26 |
| Table 36. Minimental Test: Comparison between visits and baseline | 27 |
| Table 37. Barthel Index: Results for each patient | 29 |
| Table 38. Barthel Index: Summary in each visit | 29 |
| Table 39. Barthel Index: Comparison between visits and baseline | 30 |
| Table 40. Satey results summary | 32 |
| Table 41. Frequencies of all adverse events | 32 |
| Table 42. Most frequent adverse events | 33 |
| Table 43. Most frequent adverse events with grades | 34 |
| Table 44. Frequency of Toxicities | 35 |
| Table 45. Most frequent Toxicities | 35 |
| Table 46. Most frequent Toxicities with grades | 36 |
| Table 47. List of SAEs | 37 |
| Table 48. List of all toxicities | 38 |
| Table 49. Long survivors | 38<br>41 |
| Table 50. Long survivors | 41 |
| | 41 |
| Table 51. Baseline and tumour characteristic vs long survivors | 42 |

# Figures:

DATE: 29/11/2022 (version 1.3)


### Study GEINO 13

### STATISTICAL REPORT: TABLES, LISTS AND FIGURES

Sponsor: GRUPO ESPAÑOL DE INVESTIGACIÓN EN NEUROONCOLOGÍA

| Figure 1. Progression Free Survival | 18 |
|---|---|
| Figure 2. Overall Survival | 20 |
| Figure 3. Use of corticoids | 25 |
| Figure 4. Minimental Test evolution | 28 |
| Figure 5. Barthel Index evolution | 31 |
| Figure 6. Progression Free Survival (R format) | 43 |
| Figure 7. Overall Survival (R format) | 43 |
| Figure 8. Swimmer plot: patient's follow-up | 44 |
| Figure 9. Spider plot: % change in lessions measurements from baseline | 45 |
| Figure 10. Spider plot: % change in lessions measurements from baseline ( | excluding |
| outlier value) | 45 |

DATE: 29/11/2022 (version 1.3)

### 1. RESULTS (TABLES, LISTS AND FIGURES)

The database of the study was closed on the 10-10-2019.

### 1.1. STUDY POPULATION

### 1.1.1. SCREENED PATIENTS

A total of xx patients were screened and eventually xx patients fulfilled all the inclusion and exclusion criteria.

| | Table 1. Screened patients | | |
|---|---|---|---|
| | | N | % |
| Hospital | Name | | |
| | | | - |
| | Total | | |
| Fulfils every | Patient fulfils all the inclusion criteria and none of exclusion according to the | | |
| inclusion and<br>none of the | protocol Patient does not fulfil the eligibility criteria | | |
| exclusion<br>criteria | Total | | |

**xx** patients were considered evaluable for the study and the reason for non-evaluability was screening failure in all the cases.

| | Table 2. Evaluable patie | nts | |
|----------------------|--------------------------|-----|---|
| | | N | % |
| Evaluable patients | No | | |
| | Yes | | |
| | Total | | |
| Non evaluable reason | Screening failure | | |
| | Total | • | |

Table 3. Patients included and excluded from each hospital

| | | N | О | Υ | es | To | tal |
|----------|------|---|---|---|----|----|-----|
| | | N | % | N | % | N | % |
| Hospital | Name | | | | | | |

### STATISTICAL REPORT: TABLES, LISTS AND FIGURES

Sponsor: GRUPO ESPAÑOL DE INVESTIGACIÓN EN NEUROONCOLOGÍA

Those patients excluded from the analysis are listed in the following table.

Table 4. List of patients excluded from the analysis

| Patient<br>number | Hospital | Non evaluable reason | Fulfils every inclusion and none of the exclusion criteria |
|---|---|---|---|
| 1 | | | |
| 2 | | | |
| 3 | | | |
| 4 | | | |

DATE: 29/11/2022 (version 1.3) CONFIDENTIAL


### **DEMOGRAPHIC AND CLINICAL BASELINE CHARACTERISTICS**

The median of the age was xx years and xx % were males.

| | T | able 5. A | \ge | | | | |
|---|---|---|---|---|---|---|---|
| | | N | Mean | SD | Median | Min | Max |
| Age in years (at informed conse | nt signature) | | | | | | |
| | Table 6. | Gender | and race | | | | |
| | | | N | % | | | |
| Gend | ler Men | | | | | | |
| | Femal | le | | | | | |
| | Total | | | | | | |
| Rac | e White | е | | | | | |
| | Hispar | nic | | | | | |

### 1.1.2. CLINICAL BASELINE CHARACTERISTICS

| l data |
|--------|

| | Table 7. | Clinic | cal data | | | | |
|---|---|---|---|---|---|---|---|
| | | | | N | | | % |
| Performance Status (PS) | 0<br>1<br>2<br>Total | | | | | | |
| | | N | Mean | SD | Media<br>n | Min | Max |
| Systolic blood pressure | | | | | | | |
| Diastolic blood pressure | | | | | | | |
| Weight | | | | | | | |
| Height | | | | | | | |

Table 8. Analytical data

| | N | Mean | SD | Median | Min | Max |
|------------------------|---|------|----|--------|-----|-----|
| Haemoglobin (g/dl) | | | | | | |
| Platelets (x 10e9/L) | | | | | | |
| Leukocytes (x 10e9/L) | | | | | | |
| Neutrophils (x 10e9/L) | | | | | | |
| Lymphocytes (x 10e9/L) | | | | | | |

Table 9. Biochemistry data

| | N | Mean | SD | Median | Min | Max |
|----------------------------|----------|------|----|--------|-----|-----|
| Sodium (mmol/L) | | | | | | |
| Potassium (mmol/L) | | | | | | |
| Calcium (mg/dL) | | | | | | |
| Magnesium (mg/dL) | | | | | | |
| Glucose (mg/dL) | | | | | | |
| Creatinine (mg/dL) | | | | | | |
| AST (U/L) | | | | | | |
| ALT (U/L) | | | | | | |
| Total bilirubin (mg/dL) | | | | | | |
| GGT (U/L) | | | | | | |
| Alkaline Phosphatase (U/L) | | | | | | |
| Albumin (g/dL) | | | | | | |
| LDH (U/L) | <u> </u> | | | | | |

DATE: 29/11/2022 (version 1.3) 

Table 10. Coagulation data

| Tuble 101 Gougalation auta | | | | | | |
|----------------------------|---|------|----|--------|-----|-----|
| | N | Mean | SD | Median | Min | Max |
| TP value | _ | | | | | |
| TTPA value | | | | | | |
| Fib (mg/dL) | | | | | | |
| • | | | | | | |

| Table 11. I hyroid function | | | | | | |
|-----------------------------|---|------|----|--------|-----|-----|
| | N | Mean | SD | Median | Min | Max |
| TSH value | | | | | | |
| T3 value | | | | | | |

| Table 12. ECG | |
|---------------|--------------|
| | N % |
| Qtc | Unknown |
| | <450 mseg |
| | 450-480 mseg |
| | Total |

### 1.1.3. CLINICAL TUMOUR CHARACTERISTICS

In the first surgery 16 patients (47.1%) had a tumour of grade 2 while 13 (38.2%) had a grade 3 tumour.

| iable 1 | 3. First surgery characteristics | | 0/ |
|----------------------------------|----------------------------------|---|----|
| | | N | % |
| Diagnosis with grade (First | Oligoastrocytoma grade 2 | | |
| surgery) | Oligoastrocytoma grade 3 | | |
| | Oligodendroglioma grade 2 | | |
| | Oligodendroglioma grade 3 | | |
| | Oligodendroglioma grade unknown | | |
| | Diagnosis and grade unknown | | |
| | Total | | |
| Grade (First surgery) | Grade 2 | | |
| | Grade 3 | | |
| | Unknown | | |
| | Total | | |
| Anaplasia (First surgery) | 0 | | |
| | 1 | | |
| | 2 | | |
| | 4 | | |
| | Unknown | | |
| | Total | | |
| High cellularity (First surgery) | No | | |
| | Yes | | |
| | Total | | |
| Endothelial proliferation (First | | | |
| surgery) | Yes | | |
| 3.77 | Total | | |
| Necrosis (First surgery) | No | | |
| ricordolo (i mor curgory) | Yes | | |
| | Total | | |
| Mitosis (First surgery) | No | | |
| mitosis (i list surgery) | Yes | | |
| | Total | | |
| Nuclear anomalies (First | No | | |
| surgery) | Yes | | |
| surgery) | | | |
| | Total | | |

### STATISTICAL REPORT: TABLES, LISTS AND FIGURES

Sponsor: GRUPO ESPAÑOL DE INVESTIGACIÓN EN NEUROONCOLOGÍA

Table 14. List of patients with diagnosis in first surgery

| Patie<br>numl | <br>Diagnosis with grade (First surgery) | Grade (First surgery) |
|---|---|---|
| 1 | | |
| 2 | | |
| 3 | | |
| 4 | | |
| 5 | | |

DATE: 29/11/2022 (version 1.3) 

In the last surgery, every patient (100%) was diagnosed with an oligodendroglioma grade 3.  $\,$ 

Table 15. Last surgery characteristics

| | _ | N | % |
|-------------------------------------|---------------------------|---|---|
| Diagnosis with grade (Last surgery) | Oligodendroglioma grade 3 | | |
| | Total | | |
| Grade (Last surgery) | Grade 3 | | |
| , , , , , | Total | | |
| Anaplasia (Last surgery) | 0 | | |
| | 1 | | |
| | 2 | | |
| | 3 | | |
| | 4 | | |
| | 5 | | |
| | Total | | |
| High cellularity (Last surgery) | No | | |
| | Yes | | |
| | Total | | |
| Endothelial proliferation (Last | No | | |
| surgery) | Yes | | |
| | Total | | |
| Necrosis (Last surgery) | No | | |
| | Yes | | |
| | Total | | |
| Mitosis (Last surgery) | No | | |
| | Yes | | |
| | Total | | |
| Nuclear anomalies (Last surgery) | No | | |
| | Yes | | |
| | Total | | |

### Table 16. Deletion

| | | N | % |
|--------------|-------|---|---|
| Deletion 1p | Yes | | |
| | Total | | |
| Deletion 19q | Yes | | |
| - | Total | | |

In x patients (xx%) the surgery was not completed. Biopsy was performed in x patients (xx%) and craniotomy in XX patients (xx%).

Table 17. Surgery compliance

| | | N | % |
|------------------|----------------------------------|---|---|
| Surgery | No | | |
| | Yes | | |
| | Total | | |
| Type of surgery | Biopsy | | |
| | Craniotomy | | |
| | No applicable (Surgery not done) | | |
| | Total | | |
| Relapse location | Bihemispheric | | |
| | Cingulate (right) | | |
| | (Indicate locations) | | |
| | Total | | |

The baseline barthel index mean was xx and the baseline minimental test mean was xx (data was available in xx patients).

Table 18. Baseline Barthel Index and Minimental test

| | THE STATE OF THE S | | | | | |
|---|---|---|---|---|---|---|
| | N | Mean | SD | Median | Min | Max |
| Barthel index (baseline) | | | | | | |
| Mini mental test (baseline) | | | | | | |

### 1.2.3. PREVIOUS PATHOLOGIES

For 9 patients (26.5%) previous pathologies were not reported. In those patients with previous pathologies, seizures were the most common (n=7, 17.6%) previous pathology.

Table 19. Previous pathologies

| | | N | % |
|-------------|--------------------------------------------|---|---|
| Previous | No | | |
| pathologies | Yes | | |
| | Total | | |
| | | N | % |
| Previous | .(Indicate previous pathologies. Exemples: | | |
| pathologies | Fatigue | | |
| | Cognitive disturbance | | |
| | Muscle weakness left-sided | | |

STATISTICAL REPORT: TABLES, LISTS AND FIGURES

Table 20. List of previous pathologies
Previous pathology

Sponsor: GRUPO ESPAÑOL DE INVESTIGACIÓN EN NEUROONCOLOGÍA Study GEINO 13


DATE: 29/11/2022 (version 1.3)

### 1.2. EFFICACY ANALYSES

### 1.2.1. PRIMARY EFFICACY ANALYSES: PFS

At 6 and 9 months the estimated PFS was 21.23% (with 95% CI 11-40.97), at 12 months it was 16.99% (with 95% CI 7.71-37.43) and from 18 to 48 months it was 11.32% (with 95% CI 3.68-34.86).

The median of PFS was 2.84 months (with 95% CI 2.71-5.39).

Table 22. PFS estimated survival ratio

| Progression Free Survival | Events (%, total N) | Patients at risk | % estimated cumulative<br>survival ratio | CI 95% |
|---|---|---|---|---|
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| At 18 months | | | | |
| At 24 months | | | | |
| At 30 months | | | | |
| At 36 months | | | | |
| At 42 months | | | | |
| At 48 months | | | | |

Note: Estimated using Kaplan-Meier product-limit method

Table 23. Median/mean PFS (estimated by Kaplan-Meier)

| | Median (months) | CI 95% | Mean | CI 95% |
|---------------------------|-----------------|--------|------|--------|
| Progression Free Survival | | | | |

Note: Estimated using Kaplan-Meier product-limit method

Figure 1. Progression Free Survival



In the 28 patients with PD, the median until progression was 2.8 months.

Table 24. Time until PD/exitus (only pts with event)

| Overall | Overall<br>(N=xx) |
|----------------------|-------------------|
| Time until PD/Exitus | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median (95%CI) | |
| Range | |

### 1.3.2. SECONDARY EFFICACY ANALYSES

### 1.2.2.1 OS

At 6 months the estimated OS was xx % (with xx% CI xx-xx), at 9 months it was xx % (with xx% CI xx-xx), at xx months it was ....

The median of OS was xxx months (with xx% CI xx-xx)

Table 25. OS estimated survival ratio

| Overall Survival | Events (%, total N) | Patients at risk | % estimated cumulative<br>survival ratio | CI 95% |
|---|---|---|---|---|
| At 6 months | | | | |
| At 9 months | | | | |
| At 12 months | | | | |
| At 18 months | | | | |

Note: Estimated using Kaplan-Meier product-limit method

Table 26. Median/mean OS (estimated by Kaplan-Meier)

| | Median (months) | CI 95% | Mean | CI 95% |
|------------------|-----------------|--------|------|--------|
| Overall Survival | | | | |

Note: Estimated using Kaplan-Meier product-limit method

Figure 2. Overall Survival



In those patients who died (n=xx), the median of follow-up was xx months.

Table 27. Time until exitus (only deaths)

| Overall | Overall<br>(N=xx) |
|-------------------|-------------------|
| Time until Exitus | |
| N | |
| Mean (95%CI) | |
| SD | |
| Median | |
| (95%CI) | |
| Range | |

In overall, the median of follow-up was xx months (minimum xx months and maximum of xx months).

Table 28. Time of follow-up (all patients)

| Overall | Overall (N=xx) |
|-------------------|----------------|
| Time until Exitus | |
| N | |
| Mean (95%CI) | |
| SD | |

| Overall | Overall (N=xx) |
|---------|----------------|
| Median | |
| (95%CI) | |
| Range | |

1.2.2.2 RESPONSES
13 patients (38.2%, with 95% CI 21.9-54.6), reached clinical benefit (all were Stable Disease).

Table 29. Best response and Clinical benefit rate N (%, 95% CI) Best response CR rate SD PD No evaluated Total Clinical benefit No rate Yes (CR or PR or SD) No evaluable Total

In xx patients (xx%) the reason to end of treatment was PD; xx patients (xx%) were alive at the end of follow-up.

| | | N (%) |
|---|---|---|
| Current | End of treatment due to patient decision and patient is alive at end of follow-up | |
| status | End of treatment due to PD and patient is alive at end of follow-up | |
| | End of treatment due to PD and patient is exitus | |
| | End of treatment but reason not reported and patient is exitus | |
| | End of treatment due to lack of clinical benefit and patient is alive at end of follow-up | |
| | On treatment | |
| | Total | |
| End of | PD | |
| treatment | Toxicity (with PD) | |
| reason | Patient decision | |
| | On treatment | |
| | No clinical benefit | |
| | Total | |
| Status at | Alive | |
| end of | Exitus | |
| follow-up | Total | |

**1.2.2.3 RANO EVALUATION** xx patients (xx%) presented PD in RANO evaluations, xx (xx%) of them in the 2nd RANO, x (xx%) the 3rd, x (xx%) in the 5th and x (xx%) in the 6th.

Table 31. RANO Evaluation (I)

| | | וומווים בייניים בייניים ומשו | |
|---|---|---|---|
| | | | % N |
| RANO | Without PD in RANO | | |
| <u>ō</u> | . 2 | | |
| with DD | | | |
| 1 | u co | | |
| | 9 | | |
| Reason of | 1 | | |
| PD with | T1-Gd+; T2-FLAIR: / New lesions: New appearance/ Corticoids evolution (last 5 days): Stable/ Clinical evaluation (neurological); Stable | nce/ Corticoids evolution (last 5 days): Stab | le/ Clinical evaluation (neurological): Stable |
| RANO | | | |
| | Total | | |
| DAT | DATE: 29/11/2022 (version 1.3) | CONFIDENTIAL | |

### Table 32. RANO Evaluation (II)

| | Table 32. RANO Evaluation (II) | | |
|--------------|--------------------------------|---|---|
| | | N | % |
| | NA or not reported | | |
| T1Gd+ (PD | Decrease <5% or Increase < 25% | | |
| RANO) | Increase >/= 25%* | | |
| | Total | | |
| | NA or not reported | | |
| T2/FLAIR | Increase | | |
| (PD RANO) | Stable | | |
| | Total | | |
| | NA or not reported | | |
| New lesions | New appearance | | |
| (PD RANO) | No | | |
| | Total | | |
| | NA or not reported | | |
| Corticoids | Decrease | | |
| evolution | Increase | | |
| (PD RANO) | No corticoids | | |
| (i b italio) | Stable | | |
| | Total | | |
| Clinical | NA or not reported | | |
| evaluation | Stable | | |
| (PD RANO) | Worsening | | |
| (FD RANO) | Total | | |
| | - | | |

Study GEINO 13

STATISTICAL REPORT: TABLES, LISTS AND FIGURES Sponsor: GRUPO ESPAÑOL DE INVESTIGACIÓN EN NEUROONCOLOGÍA Table 33. List of patients with RANO progressions with details Reason of PD with RANO

Patient Evaluation number RANO con PD

| | Evample: T1-Cd+:lpcroses >/- | 350/*/ T2 El AID: Stable/ New lecione: | Evample T1 (Ad-inavasca N- 250/4) T2 El AlD: Crabial Maur beinne: Mal Portionide avalution (hast E daur). No nortinaled (Tininal avaluation fraunchonias): Ctable | evaluation (neurological): Stable |
|---|---|---|---|---|
| | Example: 11-Gut: Ilici ease 71- | 23%7 12-FLAIR. Stable/ New lesions. | . INOT COTTICOTUS EVOIDITIOTI (TASE 3 DAYS). INO COTTICOTUST CITITICAL E | evaluation (neurological). Stable |
| DATE: 29/11/2022 (version 1.3) | | CONFIDENTIAL | | |

### 1.2.2.4 USE OF CORTICOIDS

x patients (xx%) reported use of corticoids.

Table 34. Use of Corticoids

| posterior decrease | | |
|--------------------|--------------------|--------------------|
| | posterior decrease | posterior decrease |

Table 35. List of patients receiving corticoids and Follow-up of dosage

| | Patient Receive | Changes in corticoids doses | C1 | C1 | C2 | C2 | C3 | C4 | C5 | C6 | C7 | C8 | C9 | C10 | C11 |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | number corticoids duri | ng from baseline (during treatment | D1 | D15 | D1 | D15 | D1 | D1 | D1 | D1 | D1 | D1 | D1 | D1 | D1 |
| | treatment (cycl | es) cycles) | | | | | | | | | | | | | |
| 7 | 1 | Evample: | | | | | | | | | | | | | |

| 1 | Yes | Example: Decreased/Increased/Stable |
|---|-----|-------------------------------------|
| 2 | | |
| 3 | | |

Figure 3. Use of corticoids



### 1.1.1.1 EVOLUTION OF MINIMENTAL TEST

The results of the minimental test for each patient (when available), is reported in the following table.

| number | <br>aı | aı | aı | αı | aı | aı | aı | ат | aı | aı | aı | aı | aı | aı | aı | aı | aı | aı | aı | aı | aı | treatment |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|

....

Patient

| Table 37. Minimenta | ıl Test: | Summary in each | visit |
|---|---|---|---|
| | N | Mean (SD) | Median (Min-Max) |
| Test Minimental (baseline) | | | |
| Test Minimental (cycle 2 d1) | | | |
| Test Minimental (cycle 3 d1) | | | |
| Test Minimental (cycle 4 d1) | | | |
| Test Minimental (cycle 5 d1) | | | |
| Test Minimental (cycle 6 d1) | | | |
| Test Minimental (cycle 7 d1) | | | |
| Test Minimental (cycle 8 d1) | | | |
| Test Minimental (cycle 9 d1) | | | |
| Test Minimental (cycle 10 d1) | | | |
| Test Minimental (cycle 12 d1) | | | |
| Test Minimental (cycle 13 d1) | | | |
| Test Minimental (cycle 14 d1) | | | |
| Test Minimental (cycle 15 d1) | | | |
| Test Minimental (cycle 16 d1) | | | |
| Test Minimental (cycle 17 d1) | | | |
| Test Minimental (cycle 18 d1) | | | |
| Test Minimental (cycle 19 d1) | | | |
| Test Minimental (cycle 20 d1) | | | |
| Test Minimental (cycle 21 d1) | | | |
| Test Minimental (cycle 22 d1) | | | |
| Test Minimental (cycle 23 d1) | | | |
| Test Minimental (end of treatment) | | · | |

.

| Table 38. Minimental Test | : Comp | <u>arison betwee</u> | n visits and baseline | |
|---|---|---|---|---|
| | N | Mean (SD) | Median (Min-Max) | p-valor <sup>1</sup> |
| Test Minimental (baseline) | | | | |
| Test Minimental (cycle 2 d1) | | | | |
| Test Minimental (baseline) | | | | |
| Test Minimental (cycle 3 d1) | | | | |
| Test Minimental (baseline) | | | | |
| Test Minimental (cycle 4 d1) | | | | |
| Test Minimental (baseline) | | | | |
| Test Minimental (cycle 5 d1) | | | | |
| Test Minimental (baseline) | | | | |
| Test Minimental (cycle 6 d1) | | | | |
| Test Minimental (baseline) | | | | |
| Test Minimental (cycle 7 d1) | | | | |
| Test Minimental (baseline) | | | | |
| Test Minimental (cycle 8 d1) | | | | |
| Test Minimental (baseline) | | | | |

DATE: 29/11/2022 (version 1.3)


Test Minimental (cycle 9 d1)
Test Minimental (baseline)
Test Minimental (cycle 10 d1)
Test Minimental (baseline)
Test Minimental (end of treatment)
1: Wilcoxon test



Figure 4. Minimental Test evolution

### 1.1.1.2 EVOLUTION OF BARTHEL INDEX

The results of the Barthel Index for each patient (when available), is reported in the following table.

| Table 40. Barthel Ind | lex: Su | mmary in each v | <i>r</i> isit |
|---|---|---|---|
| | N | Mean (SD) | Median (Min-Max) |
| Barthel Index (baseline) | | | |
| Barthel Index (cycle 2 d1) | | | |
| Barthel Index (cycle 3 d1) | | | |
| Barthel Index (cycle 4 d1) | | | |
| Barthel Index (cycle 5 d1) | | | |
| Barthel Index (cycle 6 d1) | | | |
| Barthel Index (cycle 7 d1) | | | |
| Barthel Index (cycle 8 d1) | | | |
| Barthel Index (cycle 9 d1) | | | |
| Barthel Index (cycle 10 d1) | | | |
| Barthel Index (cycle 11 d1) | | | |
| Barthel Index (cycle 12 d1) | | | |
| Barthel Index (cycle 13 d1) | | | |
| Barthel Index (cycle 14 d1) | | | |
| Barthel Index (cycle 15 d1) | | | |
| Barthel Index (cycle 16 d1) | | | |
| Barthel Index (cycle 17 d1) | | | |
| Barthel Index (cycle 18 d1) | | | |
| Barthel Index (cycle 19 d1) | | | |
| Barthel Index (cycle 20 d1) | | | |
| Barthel Index (cycle 21 d1) | | | |
| Barthel Index (cycle 22 d1) | | | |
| Barthel Index (cycle 23 d1) | | · | · |
| Barthel Index (end of treatment) | | · | |

The Barthel Index result in each visit was compared with the baseline result in those cases with results for at least 4 patients (for each pairwise comparison only those patients with measures in both visits could be compared). No statistically significant differences were found in any of the comparisons with baseline.

Table 41. Barthel Index: Comparison between visits and baseline

| | N | Mean (SD) | Median (Min-Max) | p-valor1 |
|---------------------------|---|-----------|------------------|----------|
| Barthel Index(baseline) | | | | |
| Barthel Index(cycle 2 d1) | | | | |
| Barthel Index(baseline) | | | | |
| Barthel Index(cycle 3 d1) | | | | |
| Barthel Index(baseline) | | | | |
| Barthel Index(cycle 4 d1) | | | | |
| Barthel Index(baseline) | | | | |
| Barthel Index(cycle 5 d1) | | | | |
| Barthel Index(baseline) | | | | |
| Barthel Index(cycle 6 d1) | | | | |
| Barthel Index(baseline) | | | | |
| Barthel Index(cycle 7 d1) | | | | |
| Barthel Index(baseline) | | | | |
| ` ' | | | | |

DATE: 29/11/2022 (version 1.3)


### STATISTICAL REPORT: TABLES, LISTS AND FIGURES

Sponsor: GRUPO ESPAÑOL DE INVESTIGACIÓN EN NEUROONCOLOGÍA

| Barthel Index(cycle 8 d1) |
|---------------------------------|
| Barthel Index(baseline) |
| Barthel Index(cycle 9 d1) |
| Barthel Index(baseline) |
| Barthel Index(cycle 10 d1) |
| Barthel Index(baseline) |
| Barthel Index(end of treatment) |

1: Wilcoxon test

Figure 5. Barthel Index evolution



### 1.2. SAFETY ANALYSES

Every patient but one presented at least one adverse event during follow-up (n=xx, xx%). xx patients (xx%) presented at least one adverse event grade $\geq$ 3 during follow-up. xx patients (x%) presented at least one toxicity (related AE) during follow-up. xx patients (xx%) presented at least one toxicity grade $\geq$ 3 (related AE) during follow-up. xx patients (xx%) presented at least one SAE during follow-up, and none was reported as related to the treatment.

| | | N | % |
|-----------------------|-------|---|---|
| AE | No | | |
| | Yes | | |
| | Total | | |
| Adverse event grade≥3 | No | | |
| - | Yes | | |
| | Total | | |
| Toxicity (any) | No | | |
| | Yes | | |
| | Total | | |
| Toxicity grade≥3 | No | | |
| | Yes | | |
| | Total | | |
| SAE (any) | No | | |
| | Yes | | |
| | Total | · | |
| SAE related | No | | |
| | Total | | |

### 1.2.1.

### 1.2.2. ADEVERSE EVENTS

The most frequent adverse event (any grade) were xxxxx (xx%, n=xx)....

| Table 42 | Ereguencies of all adverse events |
|----------|-----------------------------------|

| | | N | % |
|---------|----------------------------|---|---|
| Adverse | EXAMPLES: | | |
| event | Neutrophil count decreased | | |
| | Fatigue | | |
| | Platelet count decreased | | |
| | Anaemia | | |

%: calculated respect the total number of patients (N=34)

The most frequent adverse events, (at least in 10% of the patients, n=xx), are reported in the following table:

| Table 44. Most frequent adverse events | | | |
|----------------------------------------|-------|----|--------|
| | | N | % |
| Specify Adverse events. | No | 10 | 29.4% |
| EXAMPLE: Fatigue | Yes | 24 | 70.6% |
| • | Total | 34 | 100.0% |
| | No | 14 | 41.2% |
| | Yes | 20 | 58.8% |

Study GEINO 13

### STATISTICAL REPORT: TABLES, LISTS AND FIGURES

Sponsor: GRUPO ESPAÑOL DE INVESTIGACIÓN EN NEUROONCOLOGÍA

| Total | 34 | 100.0% |
|-------|----|--------|

The most frequent adverse events with their respective grades are reported in the following table:

| Table 45 Mo | st frequent adverse ( | events with grades |
|-------------|-----------------------|--------------------|

| | | No | | G1 | | G2 | | 33 | | 34 | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | % | N | % | N | % | N | % | N | % | N | % |
| Specify Adverse events. | | | | | | | | | | | | |
| EXAMPLE: Fatigue | | | | | | | | | | | | |

DATE: 29/11/2022 (version 1.3)


### 1.2.2. TOXICITIES

The most frequent toxicities (related AE of any grade) were xxx decreased (xx%, n=xx)....

### Table 46. Frequency of Toxicities

| | | N | % |
|---------|-----------------------------------------------------------|---|---|
| Adverse | Specify Advert event. EXAMPLE: Neutrophil count decreased | | |
| event | | | |
| _ | | | |

%: calculated respect the total number of patients (N=xx)

The most frequent toxicities (at least in 10% of the patients, n=x), are reported in the following table:

| Table | 47 | Most | fraguant | Toxicities |
|-------|-----|------|----------|------------|
| lable | 41. | MOSE | neaueni | TOXICILIES |

| | • | N | % |
|---------------------------|-------|---|---|
| Specify Advert event | No | | |
| EXAMPLE: Neutrophil count | Yes | | |
| decreased | Total | | |
| | No | | |
| | Yes | | |
| | Total | | |

The most frequent toxicities with their respective grades are reported in the following table:

| Table 48. Most | frequent | Toxicities | with | grades |
|----------------|----------|------------|------|--------|
|----------------|----------|------------|------|--------|

| | | No | | G1 | | G2 | ( | 33 | ( | 64 | To | otal |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | N | % | N | % | N | % | N | % | N | % | N | % |
| Specify Advert event | | | | | | | | | | | | |
| Specify Advert event<br>EXAMPLE: Neutrophil count | | | | | | | | | | | | |
| decreased | | | | | | | | | | | | |

### 1.2.3. SERIOUS ADVERSE EVENTS

| - | Table | 40 | I ict | ٠f | CA | E- |
|---|-------|----|-------|----|----|----|

| | Patient<br>number | Hospital | AE grade | Relation | Intensity | Action | SAE<br>(any) |
|---|---|---|---|---|---|---|---|
| 1 | | | | | | | |
| 2 | | | | | | | |
| 3 | | | | | | | |

DATE: 29/11/2022 (version 1.3)


### 1.3. ANNEX I: LIST OF ALL TOXICITIES

Table 50. List of all toxicities

| Patient number | Hospital | AE grade | Relation | Intensity | Action | SAE (any) |
|---|---|---|---|---|---|---|
| 1 | | | | | | |
| 2 | | | | | | |
| 3 | | | | | | |
| 4 | | | | | | |
| | | <u> </u> | | | | |

DATE: 29/11/2022 (version 1.3)


### 1.4. ANNEX II: ADDITIONAL RESULTS

In the event that the study coordinator considered evaluating the variables of a subgroup of patients (those of interest for the article), for example patients with progression free survival longer than 9 months (low survivors), some tables and graphs (PFS and OS) could be required

### 1.4.1. LONG SURVIVORS

| Table 51. Long survivors | | | |
|--------------------------|-------|---|---|
| | | N | % |
| Long | No | | |
| survivor | Yes | | |
| (PFS≥9m) | Total | | |

x patients were considered long survivors and are listed below:

List of long survivor patients (PFS≥9 months)

| Table 52. Long survivors | | | | | |
|---|---|---|---|---|---|
| | Patient<br>number | Time until<br>PD/Exitus | Progression Free<br>Survival | Time until<br>Exitus | Overall<br>survival |
| 1 | | | | | |
| 2 | | | | | |
| 3 | | | | | |
| 4 | | | | | |
| 5 | | | | | |
| 6 | | | | | |
| 7 | | | | | |


# 1.4.2. BASELINE AND TUMOUR CHARACTERISTICS VS LONG SURVIVORS

Those variables reported in table 1 of the article are reported below stratified by long survivors.

Table 53. Baseline and tumour characteristic vs. long survivors

| | Table 53. Baseline a | | | | |
|---|---|---|---|---|---|
| | | Long survivor (PFS≥9m) | | | p-value |
| | | No (n=27) | Yes (n=7) | Total (n=34) | |
| Age, mean +/-SD _ | median (range) | | | | |
| years | mean (SD) | | | | |
| Gender, n (%) | Male | | | | |
| Octidet, ii (70) | Female | | | | |
| _ | 0 | | | | |
| KPS, n (%) | 1 | | | | |
| | 2 | | | | |
| Double Index pr24 | median (range) | | | | |
| Barthel Index, n=31 — | mean (SD) | | | | |
| | median (range) | | | | |
| MMSE, n=31 — | mean (SD) | | | | |
| | Temozolomide | | | | |
| Prior treatments, n (%) | Nitrosoureas | | | | |
| _ | Radiotherapy | | | | |
| | Tumor | characteristics a | t first surgery | | |
| | | Oligoastroc | ytoma | | |
| _ | Grade 2 | | | | |
| -<br>- | Grade 3 | | | | |
| | Oligodendroglioma | | | | |
| Diagnosis, n (%) | Grade 2 | | | | |
| | Grade 3 | | | _ | |
| _ | Unknown | | | - | |
| | Not reported | | | | |
| Time from first AO<br>diagnosis to first — | median (range) | | | | |
| cycle, median<br>(range) months | mean (SD) | | | | |
| (runge) months | | | | | |

<sup>1:</sup> T-test for independent samples; 2: Mann-Whitney U test; 3: Fisher exact test.

### 1.4.3. ADDITIONAL FIGURES

### Figure 6. Progression Free Survival (R format)



Figure 7. Overall Survival (R format)



Sponsor: GRUPO ESPAÑOL DE INVESTIGACIÓN EN NEUROONCOLOGÍA Study GEINO 13



DATE: 29/11/2022 (version 1.3)


Figure 9. Spider plot: % change in lesions' measurements from baseline



Patient 04-001 had measurements that are considered outliers (too extreme) and the spider graph has been repeated excluding that patient to prevent skewing the results.

Figure 10. Spider plot: % change in lesions' measurements from baseline (excluding outlier value)

